CLINICAL TRIAL: NCT00996931
Title: A Phase II Pilot Study to Determine Efficacy and Safety of Lenalidomide (Revlimid) for Treatment of Autistic Spectrum Disorders(ASD) With Regression and Markers of Cerebrospinal Fluid Cytokine Elevation and Elevated TNF-alpha Levels
Brief Title: Efficacy and Safety of Lenalidomide for Treatment of Autistic Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sutter Medical Foundation (Other)
Responsible Party: Principal Investigator, Michael G. Chez, MD, MD, Sutter Medical Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-ASD-CHEZ-0329
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-04

CONDITIONS: Autism
Keywords: autistic spectrum disorder; lenalidomide
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — 2.5 mgs per day orally for 12 weeks
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine if lenalidomide (Revlimid®)reduces proinflammatory cytokines including TNF-alpha and may actually alter the clinical course of autism for some children.

DETAILED DESCRIPTION:
Autism currently affects 1:142 births and has no definite cause. Recent research has shown possible identifying markers in neuroglial inflammation with elevated cytokines IL-1, Il-6, and MCP-1 and elevated ratios of CSF/serum levels of TNF-alpha in patients with regressive autism.

Lenalidomide (Revlimid®) is an analogue of thalidomide. Based on the improved clinical efficacy predicted for Revlimid® in its effects on TNF-alpha and other immunomodulatory cytokines, this oral compound may prove efficacious with less toxicity compared with thalidomide.

The study will evaluate the efficacy of lenalidomide by measurement of changes in EEG, clinical global impression, Childhood Autism Rating Scale, and serum and CSF (if available) TNF-alpha at the end of the study compared with the same measurements at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autistic spectrum disorder as defined by DSM-IV criteria.
* Inflammatory CSF and serum markers with elevated level of TNF-Alfa (> 50pg/ml) or other Cytokine markers such as IL-1, IL-6 or MECP-1, or serum levels of such cytokines greater than 2X normal levels even in absence of CSF markers.

or

* Patients with interictal epiliptiform EEG changes in the absences of clinical seizures, if CSF inflammatory markers are identified.
* Patients will maintain any other baseline medications for autistic problems or EEG treatment as long as on these for prior 6-8 weeks with no dosage changes. Mentally impaired minors require a parent or legal guardian to sign the informed consent.

Exclusion Criteria:

* -Diagnosis of PPD-NOS and other autism spectrum disorders.
* Any serious medical condition, laboratory abnormality, genetic, brain, structural, or psychiatric illness that would prevent the subject from participating.
* History of neutropenia, thrombocytopenia or other types of myelosuppression or risk factors for myelosuppression.
* History or risk factors for thromboembolic events.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Current use of steroids (e.g. dexamethasone, prednisone), anthracyclines (Doxil, Adriamycin).
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Known positive for HIV or infectious hepatitis, type A, B or C or tuberculosis.

Ages: 6 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chez, MD, Principal Investigator — Sutter Medical Foundation

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: Six patients will receive oral 2.5 mg daily for 12 weeks
Period: Overall Study
Arm/Group | Lenalidomide
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Lenalidomide: Six patients will receive 2.5 mg oral daily for 12 weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in TNF-alpha Levels
Description: Change in CSF-TNF-α from baseline to 12 weeks.
Time Frame: Baseline and 12 weeks
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: mean % change
Groups:
- Lenalidomide: Six subjects received oral 2.5 mg daily for 12 weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
mean % change | 57 (25)

2. Secondary Outcome: Change in Childhood Autism Rating Scale (CARS)Value From Baseline to 6 Weeks
Description: Change in CARS value from baseline to 6 weeks. Total CARS scores range from a fifteen to 60, with a minimum score of thirty serving as the cutoff for a diagnosis of autism on the mild end of the autism spectrum.
Time Frame: Baseline and 6 weeks
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: mean change in units on scale
Groups:
- Lenalidomide: oral 25 mg daily for 12 weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
mean change in units on scale | -2.08 (1.94)

ADVERSE EVENTS:
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No